CLINICAL TRIAL: NCT01334567
Title: A Rollover Protocol to Provide Subjects From Taiwan Continued Access to Tenofovir Disoproxil Fumarate After Completing Study GS-US-174-0108
Brief Title: Rollover Protocol Continued Access to Tenofovir Disoproxil Fumarate (TDF) for Subjects in Taiwan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-174-0141
Record Dates: First submitted 2010-11-04; First posted 2011-04-13 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tenofovir DF (Experimental)
  Interventions: Drug: Tenofovir DF

INTERVENTIONS:
Drug: Tenofovir DF — Provision of tenofovir disoproxil fumarate (tenofovir DF) 300 mg tablets, as prescribed by study investigators
  Other Names: Viread®

SUMMARY:
The purpose of this study is to offer subjects from centers in Taiwan who successfully complete 168 weeks of treatment in study GS US 174-0108 access to treatment with tenofovir DF for up to three additional years (144 weeks). Subjects will be followed per local standard of care. Serious adverse events (SAEs), drug accountability and patient disposition will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

* Complete all end of study visit procedures for the GS US 174-0108 study.
* Willing and able to provide written informed consent.
* A negative pregnancy test is required for female subjects at the end of study visit (i.e., screening visit for study GS-US-174-0141) for GS US 174-0108 (unless surgically sterile or greater than two years post-menopausal)
* All sexually active female subjects who are not post menopausal, or surgically sterile and are of childbearing potential must agree to use a highly effective method of contraception during heterosexual intercourse throughout the study.
* Male subjects who are sexually active are required to use barrier contraception (condom with spermicide) during heterosexual intercourse through to study completion.

Exclusion Criteria:

• Not Applicable

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
No statistical analyses are planned. Listings will include subject enrollment, subject disposition and SAEs. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, PharmD, Study Director — Gilead Sciences
Locations (4):
- Taiwan (4):
  - Kaoshiung Hsien
  - Tainan
  - Taipei
  - Taoyuan Hsien